CLINICAL TRIAL: NCT05103254
Title: A Post-marketing, Long-term, Observational, Descriptive Study to Assess the Risk of Pregnancy and Maternal Complications and Adverse Effects on the Developing Fetus, Neonate, and Infant Among Women Exposed to Bempedoic Acid or Bempedoic Acid/Ezetimibe Fixed Combination Drug Product (FCDP) During Pregnancy
Brief Title: Bempedoic Acid Pregnancy Surveillance Program
Status: Recruiting | Type: Observational
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1002-074
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy; Hyperlipidemias
Keywords: bempedoic acid
MeSH Terms: conditions — Hyperlipidemias | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Bempedoic Acid — Bempedoic Acid 180 MG
  Other Names: Nexletol
Drug: Bempedoic Acid / Ezetimibe — Bempedoic Acid 180 MG / Ezetimibe 10 MG
  Other Names: Nexlizet

SUMMARY:
Bempedoic acid pregnancy surveillance program

DETAILED DESCRIPTION:
A surveillance study of females exposed to bempedoic acid or bempedoic acid/ezetimibe fixed combination drug product (FCDP) during pregnancy. Observational outcome data will be collected on pregnant females through pregnancy and infants through the first year of life.

ELIGIBILITY:
Inclusion Criteria:

Exposure to at least 1 dose of bempedoic acid or bempedoic acid/ezetimibe FCDP at any time during pregnancy (from first day of last menstrual period [LMP] to pregnancy outcome

Exclusion Criteria:

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Major congenital malformations (MCM) | Birth up to 12 months
  An abnormality of body structure or function that is present at birth, is of prenatal origin (i.e., birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention (CDC 2019a). MCMs will be defined and coded with criteria specified by US CDC Metropolitan Atlanta Congenital Defects Program (MACDP).

SECONDARY OUTCOMES:
Minor congenital malformation | Birth up to 12 months
  An anomaly or abnormality of body structure that is present at birth, is of prenatal origin (i.e., birth defect), poses no significant health problem in the neonatal period, and tends to have limited social or cosmetic consequences for the affected individual (CDC 2019a). The surveillance program defines and codes minor congenital malformations with criteria specified as defined by CDC (CDC 2017).
Spontaneous abortion | Time of conception up to birth
  An involuntary fetal loss or the expulsion of the products of conception occurring at < 20 gestational weeks.
Stillbirth | Time of conception up to birth
  As defined by the American College of Obstetricians and Gynecologists (ACOG), an involuntary fetal loss occurring at ≥ 20 gestational weeks or, if gestational age is unknown, a fetus weighing ≥ 350 g.
Elective termination | Time of conception up to birth
  A voluntary fetal loss or interruption of pregnancy, including pregnancy termination that occurs electively, to preserve maternal health or due to fetal abnormalities.
Preterm birth | Time of conception up to birth
  A live birth occurring at < 37 gestational weeks.
Small for gestational age (SGA) | Birth up to 12 months
  Weight at birth in < 10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants (Battaglia 1967). For the determination of SGA, the surveillance program will utilize the sex-specific international growth reference standards from the International Fetal and Newborn Growth Consortium for the 21st Century (INTERGROWTH-21st) for those born between 240/7 and 426/7 gestational weeks (Villar 2014; Villar 2016). The INTERGROWTH-21st standards are the latest available global reference standards, representing contemporary information from an international, multiethnic, diverse population, and have been specifically developed for modern research.
Postnatal growth deficiency | Birth up to 12 months
  Weight in < 10th percentile for sex and chronological age using standard growth charts. Postnatal growth deficiency will be evaluated at 4 and 12 months of infant age. For the determination of postnatal growth deficiency, the surveillance program will utilize the sex-specific international growth reference standards from the World Health Organization for children ages 0 to 24 months. The World Health Organization growth standards are recommended for use in the US for infants and children 0 to 2 years of age (CDC 2010).
Infant development deficiency | Birth up to 12 months
  Failure to achieve the developmental milestones for chronological age, as defined by the CDC (CDC 2019b). Infant developmental deficiency will be evaluated at 4 and 12 months of infant age for each CDC-defined category (social/emotional, language/communication, cognitive, and movement/physical development), separately.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Broestl, MS, Study Director — Esperion Therapuetics
Locations (1):
- Evidera, PPD business unit, Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paponja K, Pecin I, Reiner Z, Banach M. Bempedoic acid: new evidence and recommendations on use. Curr Opin Lipidol. 2024 Feb 1;35(1):41-50. doi: 10.1097/MOL.0000000000000911. Epub 2023 Dec 8. PMID 38085172